CLINICAL TRIAL: NCT07124767
Title: The Effects Of Tüber Low Insulinemic Index And Tüber Healthy Nutrition Recommendations On Overweight And Obese Patients With Polycystic Ovary Syndrome
Brief Title: The Effects Of Low Insulinemic Index Diet On Overweight And Obese Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betül Gümüş (Other)
Responsible Party: Sponsor-Investigator, Betül Gümüş, principal investigator, Atlas University
Organization: Atlas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 28.06.2024-993352
Record Dates: First submitted 2025-07-24; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: PCOS (Polycystic Ovary Syndrome); Insulinemic Response
Keywords: PCOS; Food insulinemic index; Türkiye nutrition guidelines
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet

STUDY DESIGN:
Intervention Model Description: randomized single blind two group study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tüber diet group (Active Comparator): Tüber diet group consists of 15 people. These patients of PCOS had a diet intervention according to Turkiye nutrition guidelines for 6 weeks period.
  Interventions: Other: 6 weeks of dieting according to TÜBER nutrition recommendations
- low food insulin index group (Active Comparator): low food insulin index group consists of 15 people. These patients of PCOS had a diet intervention with food selected according to their insulin indexes for 6 weeks period.
  Interventions: Other: 6 weeks of diet with low insulin index diet

INTERVENTIONS:
Other: 6 weeks of diet with low insulin index diet — 6 weeks diet period for the low insulin index group. this group has a diet programme assigned by the conductor dietitian.
  Arms: low food insulin index group
Other: 6 weeks of dieting according to TÜBER nutrition recommendations — 6 weeks of diet according to the TÜBER recomendations were applied to this group. Diets were assigned by the conductor dietitian.
  Arms: tüber diet group

SUMMARY:
The aim of this study was to investigate the relationship between PCOS and insulinemic index in overweight and/or obese women with PCOS and to evaluate potential beneficial effects on PCOS. In this study, overweight and obese women with PCOS were divided into two groups. The first group (n=15) received a 6-week nutritional program consisting of low insulin index foods as recommended by TÜBER, while the other group (n=15) received the healthy eating recommendations outlined in TÜBER. Differences in endocrine, metabolic, and anthropometric parameters between these two groups were examined after each 6-week dietary intervention.

DETAILED DESCRIPTION:
Research Type, Location, Time, and Sample Selection The aim of this randomised controlled study is to determine the effect of the food insulin index on metabolic (glucose, insulin, C-peptide) and endocrine parameters (LH, FSH, testosterone) as well as anthropometric measurements in overweight and obese women diagnosed with PCOS. In line with this objective, overweight and obese women with PCOS were divided into two groups and followed for 6 weeks; the first group (n=15) was given a diet consisting of foods with a low insulin index selected from the Turkish Nutrition Guide (TÜBER), while the other group (n=15) followed the healthy dietary recommendations outlined in TÜBER. The differences in endocrine, metabolic, and anthropometric parameters between the groups and compared to their baseline values were examined following the diets.

The study population consisted of women who were newly diagnosed with PCOS, met the inclusion criteria, and signed the informed consent form between February 2024 and February 2025 at the Atlas University Medicine Hospital's gynaecology and obstetrics clinic, following ethical committee approval. Approval for the study was obtained from the Clinical Ethics Committee of Istanbul Cerrahpaşa University, and the study was conducted in accordance with the ethical principles of the Helsinki Declaration. The purpose of the study was clearly explained to all participants, and written informed consent forms were obtained. Participants in groups 1 and 2 completed a general information form, underwent anthropometric measurements, and had their biochemical measurements recorded. Biochemical measurements obtained from patients and found in their files were transferred to the researcher's biochemical parameters form. Interviews with patients were conducted at the hospital's diet clinic.

The study was conducted with 30 overweight or obese PCOS patients. The first group, consisting of 15 patients, completed the study with a nutrition programme consisting of foods with a low insulin index according to TÜBER, while the second group, consisting of 15 patients, completed the study by applying the healthy nutrition principles specified in TÜBER.

General Plan of the Study Patients who visited the Gynaecology and Obstetrics Outpatient Clinic of Atlas University Medicine Hospital, were diagnosed with PCOS, met the inclusion criteria. Anthropometric measurements (height, waist circumference, and body composition) were taken by the researcher, and a 24-hour dietary record was recorded by a dietitian using a reminder method. The physical activity questionnaire was completed by the researcher, portion sizes of foods were explained using visuals and replicas, and biochemical parameters were obtained from patient files and processed into biochemical parameters.

Nutrition plans were prepared by the dietitian and explained to the patients based on anthropometric measurements, physical activity status, food consumption records, and biochemical parameters, and the patients were randomly assigned to a diet group (TÜBER Low Insulinemic Index and TÜBER Healthy Nutrition Recommendations) without knowing which group they were in. Patients were monitored weekly for six weeks, and they were asked to keep a 24-hour food consumption record, with macro and micro nutrient intake recorded based on the food consumption record.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese premenopausal women (BMI between 25-49.9 kg/m2),
* Being between 18-45 years of age (childbearing age),
* No underlying metabolic disease (type 2 diabetes, hypertension, undiagnosed anemia, or any other metabolic disease on a special diet).

Exclusion Criteria:

* • Pregnancy or breastfeeding within the last 6 months

  * Presence of a concomitant disease such as kidney, liver, or heart disease, gout, or hyperuricemia
  * Use of medications that affect carbohydrate metabolism (oral contraceptive pills, metformin, antiepileptics, antipsychotics, and glucocorticoids)
  * Adherence to special nutrition therapy or a hypocaloric diet in the last three months
  * Occasional or current use of medications that may affect fluid balance, including nonsteroidal anti-inflammatory drugs, diuretics, and laxatives
  * Deficiencies in biochemical parameters and inability to adhere to the diet were exclusion criteria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | From enrollment to the end of treatment at 6 weeks
  for two groups; TÜBER nutrition recommendations diet and low insulin index diet, Anthropometric measurements were evaluated, measured and compared. Anthropometric measurements used for determination of BMI kg/m^2. BMI was determined according to world health organization guides, Comparisons were made between the beginning and end of the 6-week diet periods. IBM SPSS statistics programme was used for the comparisons.
physical activity status | beginning and end of the 6-week diet periods
  for two groups; TÜBER nutrition recommendations diet and low insulin index diet, physical activity status were evaluated, measured and compared. Physical activity of participants were questioned by using the International Physical Activity Questionnaire - Short Form (IPAQ-SF), participants were classified as sedandery, normal, active. Comparisons were made between the beginning and end of the 6-week diet periods. IBM SPSS statistics programme was used for the comparisons.
food consumption | beginning and end of the 6-week diet periods.
  for two groups; TÜBER nutrition recommendations diet and low insulin index diet, food consumption records were evaluated, measured and compared. food consumption record was taken according to FAO guidelines. it was evaluated for its calories.
  Comparisons were made between the beginning and end of the 6-week diet periods. IBM SPSS statistics programme was used for the comparisons.
biochemical parameters | beginning and end of the 6-week diet periods.
  for two groups; TÜBER nutrition recommendations diet and low insulin index diet, biochemical parameters were evaluated, measured and compared. glucose and insulin scores were used to determine the HOMA IR. Comparisons were made between the beginning and end of the 6-week diet periods. IBM SPSS statistics programme was used for the comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: betül gümüş, masters, Principal Investigator — Atlas University Hospital
Locations (1):
- Atlas University Hospital, Istanbul, Bagcılar, Turkey (Türkiye)